CLINICAL TRIAL: NCT03675516
Title: The Epidemiology of Cardiovascular Disease, Haematological Abnormalities, and Other Comorbidities in Early Rheumatoid Arthritis in the United Kingdom and Their Associations With Important Outcomes
Brief Title: Comorbidities and Outcomes in Early Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Momentum Data (Industry)
Responsible Party: Sponsor
Other Study IDs: P001
Record Dates: First submitted 2018-09-14; First posted 2018-09-18 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis cases: New onset cases of rheumatoid arthritis
  Interventions: Other: No specific intervention
- Controls: Age, gender and primary care practice-matched controls
  Interventions: Other: No specific intervention

INTERVENTIONS:
Other: No specific intervention — Usual care

SUMMARY:
Identify the burden of comorbidity at the time of diagnosis of rheumatoid arthritis. Identify the impact of comorbidity present at diagnosis on cardiovascular disease, death, rheumatoid arthritis disease progression and infections.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis prior to 1st January 2017
* Aged ≥18 years old

Exclusion Criteria:

* Patients with another other rheumatic disease

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed rheumatoid arthritis identified from their primary care records.
Sampling Method: Non-Probability Sample
Enrollment: 13182 (Actual)
Dates: Start 2004-03-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy McGovern, BSc, Study Director — Momentum Data
Locations (1):
- Momentum Data Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual patient data is confidential but can be made available in an anonymised form to bone fide researchers subject to the required data protection training and other requirements. All data will remain behind a firewall and will only be available for access through a secured computer network.

REFERENCES:
- [Result] Nikiphorou E, de Lusignan S, Mallen CD, Khavandi K, Bedarida G, Buckley CD, Galloway J, Raza K. Cardiovascular risk factors and outcomes in early rheumatoid arthritis: a population-based study. Heart. 2020 Oct;106(20):1566-1572. doi: 10.1136/heartjnl-2019-316193. Epub 2020 Mar 24. PMID 32209618
- [Result] Nikiphorou E, de Lusignan S, Mallen C, Roberts J, Khavandi K, Bedarida G, Buckley CD, Galloway J, Raza K. Prognostic value of comorbidity indices and lung diseases in early rheumatoid arthritis: a UK population-based study. Rheumatology (Oxford). 2020 Jun 1;59(6):1296-1305. doi: 10.1093/rheumatology/kez409. PMID 31580449
- [Result] Nikiphorou E, de Lusignan S, Mallen C, Khavandi K, Roberts J, Buckley CD, Galloway J, Raza K. Haematological abnormalities in new-onset rheumatoid arthritis and risk of common infections: a population-based study. Rheumatology (Oxford). 2020 May 1;59(5):997-1005. doi: 10.1093/rheumatology/kez344. PMID 31501866

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rheumatoid Arthritis Cases | Controls
Started | 6591 | 6591
Completed | 6591 | 6591
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis Cases | Controls | Total
Number analyzed (Participants) | 6591 | 6591 | 13182
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (15.8) | 59.8 (15.8) | 59.8 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4449 | 4449 | 8898
  Male | 2142 | 2142 | 4284
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4883 | 4428 | 9311
  Asian | 255 | 174 | 429
  Black | 128 | 125 | 253
  Mixed | 26 | 24 | 50
  Other | 36 | 21 | 57
  Missing | 1263 | 1819 | 3082
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6591 | 6591 | 13182

OUTCOME MEASURES:

1. Primary Outcome: Event Rate for a Cardiovascular Composite of Incident Myocardial Infarction, Stroke, or Heart Failure
Time Frame: From the date of rheumatoid arthritis diagnosis (after 1st January 2004) to the date of diagnosis of myocardial infarction, stroke, or heart failure (whichever came first) or to loss to follow-up or until 1st January 2017 (maximum follow-up: 13 years).
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Rheumatoid Arthritis Cases | Controls
Number analyzed (Participants) | 6591 | 6591
Events per 1000 person years | 10.62 [9.61 to 11.69] | 8.13 [4.26 to 9.07]

2. Primary Outcome: Event Rate for a Composite of Incident Infections.
Description: The composite will comprise incident upper respiratory tract infections, bronchitis, influenza-like illnesses, pneumonia, intestinal infectious diseases, herpes simplex, skin and soft tissue infections, urinary tract infections, and genital and perineal infections
Time Frame: From the date of rheumatoid arthritis diagnosis (after 1st January 2004) to the date of infection or to loss to follow-up or until 1st January 2017 (maximum follow-up: 13 years).
Population: This outcome was not assessed in controls
Measure: Count of Participants; unit: Participants
Arm/Group | Rheumatoid Arthritis Cases | Controls
Number analyzed (Participants) | 6591 | 0
Participants | 3506 | 0

3. Secondary Outcome: Event Rate for Incident Stroke
Time Frame: From the date of rheumatoid arthritis diagnosis (after 1st January 2004) to the date of diagnosis of stroke or to loss to follow-up or until 1st January 2017 (maximum follow-up: 13 years).
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Rheumatoid Arthritis Cases | Controls
Number analyzed (Participants) | 6591 | 6591
Events per 1000 person years | 4.29 [3.67 to 4.99] | 3.82 [3.24 to 4.48]

4. Secondary Outcome: Event Rate for Incident Heart Failure
Time Frame: From the date of rheumatoid arthritis diagnosis (after 1st January 2004) to the date of diagnosis of heart failure or to loss to follow-up or until 1st January 2017 (maximum follow-up: 13 years).
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Rheumatoid Arthritis Cases | Controls
Number analyzed (Participants) | 6591 | 6591
Events per 1000 person years | 3.98 [3.39 to 4.65] | 2.72 [2.23 to 3.29]

5. Secondary Outcome: Event Rate for a Joint Operations Composite, Comprised of Incident Joint Operations on Shoulder, Elbow, Wrist, Hand, Hip, Knee, Ankle and Foot
Time Frame: From the date of rheumatoid arthritis diagnosis (after 1st January 2004) to the date of joint operation to follow-up or until 1st January 2017 (maximum follow-up: 13 years).
Population: A comparison with controls was not included for this endpoint as this end point was only relevant to people with rheumatoid arthritis (as a marker of disease severity) and was not collected for controls.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Rheumatoid Arthritis Cases | Controls
Number analyzed (Participants) | 6591 | 0
Events per 1000 person years | 20.11 [18.63 to 21.69] |

ADVERSE EVENTS:
Time Frame: Over the follow-up period (maximum 10 years) from diagnosis to the first of: loss to follow-up, death, deregistration from care provider, or the end of the study period (1st January 2018)
Description: As there was no intervention (this was an observational study) data on adverse events was not applicable therefore All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Rheumatoid Arthritis Cases | Controls
All-Cause Mortality (participants affected / at risk) | 0/6591 | 0/6591
Serious Adverse Events (participants affected / at risk) | 0/6591 | 0/6591
Other Adverse Events (participants affected / at risk) | 0/6591 | 0/6591

LIMITATIONS AND CAVEATS:
No data was available on mortality - this outcome was therefore dropped from the analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No